CLINICAL TRIAL: NCT03607708
Title: Alternative Treatments To Prevent Cognitive Decline in Older Adults With Depression and Anxiety
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Soham Rej MD, MSc, MD, MSc, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LadyDI
Record Dates: First submitted 2018-07-11; First posted 2018-07-31 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-04

CONDITIONS: Depression Anxiety Disorder
MeSH Terms: interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness-Based Cognitive Therapy (MBCT) (Experimental): The MBCT intervention will consist of group conducted meditative practices, lasting 2 hours per week for 8 weeks. Patients will be invited to try various techniques during sessions (brief silent meditations, guided meditations, body scans, gentle arm movement exercises).
  Interventions: Other: Mindfulness-Based Cognitive Therapy (MBCT)
- Health Enhancement Program (HEP) (Active Comparator): Health Enhancement Program (HEP) : Has been previously designed and used for the purpose of being a manualized active control in meditation-based intervention trials, controlling for several non-specific factors found in a mindfulness meditation group. Participants will learn about health promotion, healthy diet, music, exercise as well as implementing positive health-enhancing life changes both in-session and during at-home practice with the support of a group facilitator, but do not learn mindfulness techniques.
  Interventions: Other: Health Enhancement Program (HEP)

INTERVENTIONS:
Other: Mindfulness-Based Cognitive Therapy (MBCT) — The MBCT intervention will consist of group conducted meditative practices, lasting 2 hours per week for 8 weeks. Patients will be invited to try various techniques during sessions (brief silent meditations, guided meditations, body scans, gentle arm movement exercises).
  Arms: Mindfulness-Based Cognitive Therapy (MBCT)
Other: Health Enhancement Program (HEP) — Health Enhancement Program (HEP) : Has been previously designed and used for the purpose of being a manualized active control in meditation-based intervention trials, controlling for several non-specific factors found in a mindfulness meditation group. Participants will learn about health promotion, healthy diet, music, exercise as well as implementing positive health-enhancing life changes both in-session and during at-home practice with the support of a group facilitator, but do not learn mindfulness techniques.
  Arms: Health Enhancement Program (HEP)

SUMMARY:
Major depression and anxiety disorders are leading causes of disability worldwide. These mental disorders deeply impact social functioning and physical health in more than 300,000-600,000 Canadians over the age of 60. Depressed and anxious older adults have a 2-3 times increased risk of developing dementia and cognitive decline.

Mindfulness-based cognitive therapy (MBCT) is a group meditation intervention that has been beneficial in treating depression and anxiety in younger adults. Our research group has experience conducting clinical trials of MBCT in older adults with depression and anxiety. Meditation therapies may prevent cognitive decline, but no previous study has examined this with MBCT.

In this 8-week clinical trial, Investigators are examining whether MBCT can strengthen the structural and functional integrity of brain networks and improve cognitive resilience in vulnerable depressed and anxious older adults. Investigators will also examine whether MBCT can improve depression, anxiety symptoms, disability, and quality of life in patients.

Investigators will conduct a pilot randomized controlled trial (RCT), comparing Mindfulness-Based Cognitive Therapy (MBCT; n=15) versus a Health Enhancement Program (HEP; n=15) active control in 30 older patients (>60) with depression or anxiety. Participants will be blinded to the treatment hypothesis while investigators and raters will be additionally blinded to group assignment. Both MBCT and HEP will be taught in weekly sessions over 8 weeks in similar sized groups (4-10 participants).

Investigators will measure the effect of these interventions on brain network function and structure using magnetic resonance imaging at baseline and 8-week timepoints. Investigators will also assess cognitive functioning and a range of clinical symptoms/quality of life measures at baseline, 8-week and 6-month follow-up.

Investigators anticipate that this project will improve quality of life in depressed and anxious older adults by enhancing brain resilience, cognitive function, and general mental health. This project will provides essential pilot data for a longer-term definitive neuroimaging trial of MBCT to assess the potential of this intervention to prevent cognitive decline and dementia in older adults.

DETAILED DESCRIPTION:
Context - Review of Literature

Depression and anxiety are common in older adults affecting 300,000-600,000 Canadian seniors annually1. About 30% of patients aged ≥60 suffering from these conditions have cognitive dysfunction across several domains 2,3, and an episode of depression or anxiety in this population increases the odds of developing dementia by two-fold4-6. Cognitive impairment and dementia are major causes of disability and dependency among older people worldwide. These conditions confer poor quality of life and place people in an extremely vulnerable condition7.

Adequate treatment of a depressive/anxiety episode can improve short- and longer-term cognition in executive, language, memory, and processing speed domains8. Because depression and anxiety in late-life are reversible to a certain extent and they are important risk factors for subsequent cognitive decline; improving these conditions can ultimately improve quality of life, lengthen the independent living of vulnerable people, reduces stress and caregiver burden. Unfortunately, existing pharmacotherapy treatments for late-life depression and anxiety have limited effectiveness (50-60% of patients are treatment-resistant), are poorly tolerated, and access is difficult due to the absence of trained personnel. Additionally, there are long waiting lists (up to 12 months) in most Canadian provinces and interventions are administered one-on-one, which is costly for the health system9. Thus, there is an urgent need for novel treatments for late-life depression and anxiety that can also improve cognition and even potentially prevent dementia in the longer-term.

Mindfulness-based cognitive therapy (MBCT) is a group intervention that teaches mindfulness meditation (non-judgemental awareness of the present moment)10. MBCT is scalable, accessible, cost efficient, and has been shown to decrease symptoms of depression, anxiety and other psychiatric disorders11. Additionally, MBCT is associated with improved quality of life 12, disability, caregiver burden and stress13. Studies conducted by our own group have found that mindfulness meditation is feasible and well-tolerated in older patients suffering from depression and anxiety14. While the neural mechanisms of MBCT are not fully understood, previous work in younger adults has shown that this intervention increases grey matter density in the brain's hippocampus, known to be involved in learning, memory and stress15. Moreover, long-term meditation practitioners displayed decreased age-related degeneration of the hippocampus16 These findings are relevant because decreased hippocampal volume17,18 and brain functional connectivity (default mode network)19 are commonly found in depressed patients. Additionally, these findings are also observed early in Alzheimer's disease and are associated with cognitive decline20.

Study Purpose and Rationale

Despite all this evidence, it remains unknown whether MBCT can strengthen brain networks, increase brain volume, and bolster cognition in depressed and anxious older adults. To our knowledge, previous mindfulness studies assessing cognition in older adults have not used MBCT nor have used neuroimaging techniques in depressed and anxious participants. Cognitive assessments in previous studies were not sensitive enough and did not use an appropriate active control group.

Thus, to address these issues, Investigators will conduct a randomized controlled trial (RCT) in late-life depression and anxiety using a standardized MBCT intervention, an appropriate active control group, a more sensitive neurocognitive test battery and the use of neuroimaging methods. In this pilot neuroimaging study, Investigators wish to assess the effects of a standard Mindfulness-Based Cognitive Therapy (MBCT) compared to an active control, Health Enhancement Program (HEP), on a number of clinical and biologically relevant outcomes, with a focus on structural and functional integrity of the default-mode network.

ELIGIBILITY:
Inclusion criteria

1. Patients will be >60 years of age presenting with clinically meaningful symptoms of depression or anxiety (PHQ-9 or GAD-7 scores ≥10).
2. Participants will be willing and able to attend at least 75% of weekly HEP or MBCT sessions.
3. Have sufficient hearing to follow verbal instructions;
4. Have adequate understanding of English and/or French.
5. Able to sit for 20-25 minutes without discomfort.

Exclusion criteria

1. Inability to provide informed consent.
2. Clinical evidence of dementia as defined by the Mini-Cog; a lifetime diagnosis of bipolar I or II disorder or primary psychotic disorder (schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder).
3. High acute risk of suicide (e.g., active suicidal ideation and/or current/recent intent or plan).
4. Severe personality disorder, that will interfere with their ability to function in a group setting.
5. Active substance use; non-correctable.
6. Clinically significant sensory impairment.
7. Diagnosed Intellectual Deficiency (e.g. Childhood Mental Retardation, Autism)
8. Acutely unstable medical illnesses, including delirium or acute cerebrovascular or cardiovascular events within the last 6 months; having a terminal medical diagnosis with prognosis of less than 12 months.
9. Currently practicing any form of meditation on a regular basis.
10. Unwilling to remain on the same psychotropic medications including dosage for the first 8 weeks of the study

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Changes in functional connectivity (rs-fMRI) from baseline to 8- week follow -up | Baseline and 8 weeks
  Using an 8- week RCT, assess the effects of MBCT (compared to an active control condition) on functional integrity of key default- mode network (DMN) nodes using functional connectivity measured by resting-state fMRI,
  Hypothesis . Compared to HEP controls, MBCT- treated patients will show larger increases from baseline to 8- week follow -up in 1) functional connectivity between regions implicated in the DMN
Structural Volume Change using structural sMRI from baseline to 8- week follow -up | Baseline and 8 weeks
  Using an 8- week RCT, assess the effects of MBCT (compared to an active control condition) on changes in changes Structural Volume
  Investigators hypothesis : Compared to HEP controls, MBCT- treated patients will show volume increase from baseline to 8- week follow -up in the bilateral hippocampal and posterior cingulate cortex nodes of the DMN,
Changes in Glutathione measured by magnetic resonance spectroscopy(MRS) from baseline to 8- week follow -up | Baseline and 8 weeks
  Increase in levels of Glutathione from baseline to 8- week follow -up in key mood regulating brain areas of the DMN (ventro-medial prefrontal cortex).

SECONDARY OUTCOMES:
Improvements in cognitive functio | Baseline and 8 weeks
  Using a 8-week RCT, assess whether MBCT is associated with improvements in cognitive function (better attention and processing speed) at 8-week follow-up. Hypothesis 2 . Compared to HEP controls, MBCT-treated patients will show greater improvements on the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) from baseline to 8-week follow-up.

OTHER OUTCOMES:
Improvements in patient depression (PHQ-9) | Baseline, 8 weeks and 26 -week follow-up
  To investigate whether MBCT is associated with improvements in patient depression (PHQ-9), compared to HEP.
  Hypothesis : MBCT will be superior to HEP at 8 week followup on depression improvement
Improvement in Cognition 26- week follow-up. | 26 -week follow-up
  To investigate the effects of MBCT and HEP on cognition at 26 -week follow-up. Hypothesis . MBCT will continue to be superior to HEP at 26 -week follow-up with regard to RBANS and all measures listed in exploratory Objective 1.
changes in Blood inflammation markers from baseline to 8 weeks | Baseline and 8 weeks
  To explore whether blood inflammation markers, predict treatment response with MBCT.
  Hypothesis 5. Depression and anxiety symptoms will be associated with levels of inflammatory markers. Levels of inflammatory markers will be decreased, in the MBCT participants at 8 -week follow-up compared to HEP, which in -turn will be associated with greater reductions in depression/anxiety scores.
Anxiety (GAD-7) | Baseline, 8 weeks and 26 -week follow-up
  To investigate whether MBCT is associated with improvements in patient Anxiety (GAD-7), compared to HEP.
  Hypothesis : MBCT will be superior to HEP at 8 week followup on Anxiety improvement
Disability (WHODAS2) | Baseline, 8 weeks and 26 -week follow-up
  To investigate whether MBCT is associated with improvements in patient Disability (WHODAS2), compared to HEP.
  Hypothesis : MBCT will be superior to HEP at 8 week followup on Disability (WHODAS2) improvement
improvement in Sleep (Athens Insomnia scale) | Baseline, 8 weeks and 26 -week follow-up
  To investigate whether MBCT is associated with improvements in patient Sleep (Athens Insomnia scale), compared to HEP.
  Hypothesis : MBCT will be superior to HEP at 8 week followup on Sleep (Athens Insomnia scale)improvement
  The Athens Insomnia scale( AIS ) was developed to assess the severity of insomnia based on the ICD-10 diagnostic criteria. It is a self-reported questionnaire consisting of 8 items; the first 5 items assess difficulty with sleep induction, awakening during the night,early morning awakening, total sleep time, and overall quality of sleep, while the last 3 items pertain to the sense of well-being,overall functioning and sleepiness during the day The usual time frame for responding is the last month. Each item of AIS can be rated 0-3, with 0 corresponding to no problem at all and 3 to very serious problem
Quality of life (Euro-QOL) | Baseline, 8 weeks and 26 -week follow-up
  To investigate whether MBCT is associated with improvements in patient Quality of life (Euro-QOL), compared to HEP.
  Hypothesis : MBCT will be superior to HEP at 8 week followup on Quality of life (Euro-QOL) improvement
Geriatric Anxiety Inventory (GAI) | Baseline, 8 weeks and 26 -week follow-up
  To investigate whether MBCT is associated with improvements in patient Geriatric Anxiety Inventory (GAI), compared to HEP.
  Hypothesis : MBCT will be superior to HEP at 8 week followup onGeriatric Anxiety Inventory (GAI) improvement

CONTACTS AND LOCATIONS:
Overall Officials: Soham Rej, MD/MSc, Principal Investigator — Lady David Institute
Locations (2):
- Canada (2):
  - Lady David Institute, Montreal, Quebec
  - Douglas Mental Health University Institute, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thomas Z, Novak M, Platas SGT, Gautier M, Holgin AP, Fox R, Segal M, Looper KJ, Lipman M, Selchen S, Mucsi I, Herrmann N, Rej S. Brief Mindfulness Meditation for Depression and Anxiety Symptoms in Patients Undergoing Hemodialysis: A Pilot Feasibility Study. Clin J Am Soc Nephrol. 2017 Dec 7;12(12):2008-2015. doi: 10.2215/CJN.03900417. Epub 2017 Oct 12. PMID 29025788
- See also: Related Info — http://geriparty.com